CLINICAL TRIAL: NCT01961258
Title: "SEVERE ASTHMA" in the COMMUNITY: How Severe it Really is and to What Extent Its Management Has Been Exhausted
Brief Title: "SEVERE ASTHMA" in the COMMUNITY
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 0016-13-MMC
Record Dates: First submitted 2013-10-07; First posted 2013-10-11 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2013-10

CONDITIONS: Severe Asthma
Keywords: Severe Asthma, Community, comorbidities, patient compliance,PFT, anti-IgE therapy
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Sever asthmatics in the comminity: Computerized data base analysis and sampling of patients for outpatient clinic evaluation.
  Interventions: Other: Computerized data base analysis and sampling of patients for outpatient clinic evaluation

INTERVENTIONS:
Other: Computerized data base analysis and sampling of patients for outpatient clinic evaluation

SUMMARY:
SEVERE ASTHMA IN THE COMMUNITY-

BACKGROUND Severe asthma is a common problem. In the world approximately 300 million people have asthma but it is estimated that only 5% of these patients have severe asthma. Although "severe asthma" comprises a small fraction of the entire asthmatic population its share in the total economic burden of asthma is 80 percent. In Israel the prevalence of asthma among adult patients is about 5-6% but the prevalence of severe asthma is unknown.

The definition of severe asthma has been changed during the years. Most recently in 2009 the WHO agreed on a unified definition of "severe asthma" that would fit countries of different socioeconomic development [1]. Severe asthma includes now 3 different groups: group one "untreated severe asthma", group two "difficult to treat severe asthma" and group three "treatment-resistant severe asthma". As all asthmatic patients in Israel have easy access to medical care, the current study will deal with the last two groups ("difficult to treat asthma" and "treatment resistant asthma").

AIMS Primary endpoints:

1. To identify the prevalence of severe asthma in the community according to the WHO definition of group two & three.
2. To assess whether anti-IgE therapy (Omalizumab), was considered in these groups of severe asthma.

Secondary endpoints:

1. To assess factors involved in "difficult to treat asthma" according to the WHO definition. Factors as patient compliance, presence of co-morbidities, symptoms of untreated potential asthma triggers including GE reflux, post nasal drip/atopic rhino-sinusitis, and intervening medications including NSAID and beta-blockers.
2. To asses the level of asthma control, level of patient follow-up care including asthma specialist visits, periodic PFT's and asthma education.
3. To assess the fraction of patients with severe asthma that is eligible to anti-IgE therapy according to the indications of the Israeli Ministry of Health (proven asthma, uncontrolled by high dose of combined ICS+LABA inhaler therapy + at least 2 courses of systemic corticosteroids in the last year + proven atopy to at least one perennial aeroallergen + IgE level of 30-1,500 IU/ml)

DESIGN A prospective non-blinded non-randomized observation study among the population insured by Clalit Medical Services (CMS) in the Sharon- Shomron Medical District in Israel.

DETAILED DESCRIPTION:
SEVERE ASTHMA IN THE COMMUNITY- STUDY PROTOCOL-SYNOPSIS

TITLE Severe Asthma in the Community: How severe it really is and to what extent its management has been exhausted PI Shabtai Varsano M.D. Head Asthma Clinic, Head-deputy Dept. of Pulmonary Medicine.

Co-investigators Shitrit David M.D, Head Dept. of Pulmonary Medicine David Segev M.D Sharon -Shomron Medical District Headquarters, Clalit Medical Services.

SITE Asthma Care & Education Unit, Dept of Pulmonary Medicine, Sapir Medical Center, Meir General Hospital Kfar-Sava, Israel.

BACKGROUND Severe asthma is a common problem. In the world approximately 300 million people have asthma but it is estimated that only 5% of these patients have severe asthma. Although "severe asthma" comprises a small fraction of the entire asthmatic population its share in the total economic burden of asthma is 80 percent. In Israel the prevalence of asthma among adult patients is about 5-6% but the prevalence of severe asthma is unknown.

The definition of severe asthma has been changed during the years. Most recently in 2009 the WHO agreed on a unified definition of "severe asthma" that would fit countries of different socioeconomic development [1]. Severe asthma includes now 3 different groups: group one "untreated severe asthma", group two "difficult to treat severe asthma" and group three "treatment-resistant severe asthma". As all asthmatic patients in Israel have easy access to medical care, the current study will deal with the last two groups ("difficult to treat asthma" and "treatment resistant asthma").

AIMS Primary endpoints:

1. To identify the prevalence of severe asthma in the community according to the WHO definition of group two & three.
2. To assess whether anti-IgE therapy (Omalizumab), was considered in these groups of severe asthma.

Secondary endpoints:

1. To assess factors involved in "difficult to treat asthma" according to the WHO definition. Factors as patient compliance, presence of co-morbidities, symptoms of untreated potential asthma triggers including GE reflux, post nasal drip/atopic rhino-sinusitis, and intervening medications including NSAID and beta-blockers.
2. To asses the level of asthma control, level of patient follow-up care including asthma specialist visits, periodic PFT's and asthma education.
3. To assess the fraction of patients with severe asthma that is eligible to anti-IgE therapy according to the indications of the Israeli Ministry of Health (proven asthma, uncontrolled by high dose of combined ICS+LABA inhaler therapy + at least 2 courses of systemic corticosteroids in the last year + proven atopy to at least one perennial aeroallergen + IgE level of 30-1,500 IU/ml)

DESIGN:

A prospective non-blinded non-randomized observation study among the population insured by Clalit Medical Services (CMS) in the Sharon- Shomron Medical District in Israel.

PROTOCOL:

The study will include all patients at the age interval of 20-70 years with bronchial asthma treated by CMS, Sharon-Shomron district. The total population at this age interval that is insured by CMS in this district is 347,374.

A. Screening of the computerized database of CMS to detect all patients at the age interval of 20-70 years with a computerized title-diagnosis of bronchial asthma during the period of January 1st -December 31, 2011. (preliminary data shows that the total asthmatic population at this age interval is 20,651 patients (5.94% of the entire population).

B. To detect from this database the asthmatic patients that are considered to have "severe asthma" according to the level of medication that is prescribed to them (adjusted on the basis of severe/refractory asthma definition by the ATS workshop consensus 2000) [2].

C. To detect the fraction of patients having co-morbidities and/or potential triggers (computerized title-diagnosis) that may interfere with asthma management (WHO group two: potentially "difficult to treat severe asthma"). Severe asthmatics without these co-morbidities /triggers will be considered as having WHO group three "treatment resistant severe asthma".

D. To detect the fraction of the patients with "severe asthma" that underwent evaluation for anti IgE-therapy.

E. To evaluate a sample of the above "severe asthma" population (WHO groups two and three) in the asthma outpatient clinic in Meir Hospital (estimated on the basis of preliminary data, 200-250 patients). If the absolute number of patients in either WHO group two or group three will not exceed 150, all patients will be invited. If the number will exceed 150, then each second patient, consecutively according to the computerized list, will be invited.

F. Patients invited to the asthma outpatient clinic will be evaluated by a pulmonary physician and complete a specific questionnaire regarding asthma control level (including non-scheduled use of medical resources), medication adherence, co-morbidities, smoking history, potential asthma triggers, level of asthma education, quality of follow-up care and potential adverse events in patients receiving anti-IgE therapy that are possibly related to this specific therapy.

G. All patients will undergo post bronchodilator spirometric evaluation, assessment of blood cell counts for peripheral eosinophils, total IgE blood levels and skin testing for aeroallergens.

H. Stages F and G of this protocol will be accomplished in one visit and there will be no more outpatint visits under this study.

Inclusion criteria:

A. Age 20-70 years old

B. A computerized diagnosis-title of "bronchial asthma", at any stage of severity. A subgroup of the above asthmatic patients will be considered as having "severe asthma" according to the ATS workshop consensus definition of severe/refractory asthma, based on the level of prescribed medication criteria 2000:

C. An obligatory criteria of at least 12 month inhaler-therapy prescription of a combination of high dose corticosteroid +LABA (at least 12 inhalers of Symbicort 160/4.5 mcg OR at least 10 inhalers of Seretide 500 mcg, a year) PLUS at least one of the following criteria:

D. Prescription of SABA, either Ventolin OR Bricalin inhalers at least once a quarter of a year or at least 4 inhalers in 12 months OR at least one prescription a month of inhalation-solution of Ventolin or Bricalin a month.

E. Prescription of an oral or IM corticosteroid, at least twice in the last 12 months.

The fulfilment of the above mentioned criteria indicates that these asthmatic patients are not conrolled, according to the GINA definition of controlled asthma.

Asthmatics that potentially have "difficult to treat severe asthma" due to co-morbidities or potential triggering factors will be sub-grouped according to these criteria (criteria for potential exclusion of having "treatment resistant severe asthma"):

A. Having computerized title-diagnosis of COPD, congestive heart failure, smoking, bronchiectasis, interstitial lung disease.

B. Prescription of an oral or topical (ocular) beta-blockers.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-70 years old
* A computerized diagnosis-title of "bronchial asthma", at any stage of severity.

A subgroup of the above asthmatic patients will be considered as having "severe asthma" according to the ATS workshop consensus definition of severe/refractory asthma, based on the level of prescribed medication criteria 2000:

- An obligatory criteria of at least 12 month inhaler-therapy prescription of a combination of high dose corticosteroid +LABA (at least 12 inhalers of Symbicort 160/4.5 mcg OR at least 10 inhalers of Seretide 500 mcg, a year)

PLUS at least one of the following criteria:

* Prescription of SABA, either Ventolin OR Bricalin inhalers at least once a quarter of a year or at least 4 inhalers in 12 months OR at least one prescription a month of inhalation-solution of Ventolin or Bricalin a month.
* Prescription of an oral or IM corticosteroid, at least twice in the last 12 months.

The fulfilment of the above mentioned criteria indicates that these asthmatic patients are not conrolled, according to the GINA definition of controlled asthma.

Asthmatics that potentially have "difficult to treat severe asthma" due to co-morbidities or potential triggering factors will be sub-grouped according to these criteria (criteria for potential exclusion of having "treatment resistant severe asthma"):

* Having computerized title-diagnosis of COPD, congestive heart failure, smoking, bronchiectasis, interstitial lung disease.
* Prescription of an oral or topical (ocular) beta-blockers.

Exclusion Criteria:

* Age <20 or >70 years old.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include all patients at the age interval of 20-70 years with bronchial asthma treated by CMS, Sharon-Shomron district.
  A. Screening of the computerized database of CMS to detect all patients at the age interval of 20-70 years with a computerized title-diagnosis of bronchial asthma during the period of January 1st -December 31, 2011, and January 1st -December 31, 2012. To detect from this database the asthmatic patients that are considered to have "severe asthma" according to the level of medication that is prescribed to them.
  B. Patients having co-morbidities and/or potential triggers (computerized title-diagnosis) that may interfere with asthma management (WHO group two: potentially "difficult to treat severe asthma"). Severe asthmatics without these co-morbidities /triggers will be considered as having WHO group three "treatment resistant severe asthma".
  C. Patients with "severe asthma" that underwent evaluation for anti IgE-therapy.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2015-06; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
The prevalence of severe asthma in the community according to the WHO definition of group two & three. | 1 year
  To identify the prevalence of severe asthma in the community according to the WHO definition of group two & three.
The prevalence of severe asthma in the community according to the WHO definition of group two & three. | 1 year
  To assess whether anti-IgE therapy (Omalizumab), was considered in these groups of severe asthma.

SECONDARY OUTCOMES:
Factors involved in "difficult to treat asthma" according to the WHO definition. | 1 year
  To assess factors involved in "difficult to treat asthma" according to the WHO definition. Factors as patient compliance, presence of co-morbidities, symptoms of untreated potential asthma triggers including GE reflux, post nasal drip/atopic rhino-sinusitis, and intervening medications including NSAID and beta-blockers.
Factors involved in "difficult to treat asthma" according to the WHO definition. | 1 year.
  To assess the level of asthma control, level of patient follow-up care including asthma specialist visits, periodic PFT's and asthma education.
Factors involved in "difficult to treat asthma" according to the WHO definition. | 1 year.
  To assess the fraction of patients with severe asthma that is eligible to anti-IgE therapy according to the indications of the Israeli Ministry of Health (proven asthma, uncontrolled by high dose of combined ICS+LABA inhaler therapy + at least 2 courses of systemic corticosteroids in the last year + proven atopy to at least one perennial aeroallergen + IgE level of 30-1,500 IU/ml)

CONTACTS AND LOCATIONS:
Overall Officials: Shabtai Varsano, M.D., Principal Investigator — Head-Deputy Dept. of Pulmonary medicine. Head of Asthma Care and Education unit.

REFERENCES:
- [Derived] Varsano S, Israeli L, Shitrit D. "Severe-controlled" asthma 4 years later: is it still controlled? J Asthma. 2021 Aug;58(8):1102-1110. doi: 10.1080/02770903.2020.1753208. Epub 2020 Apr 27. PMID 32338094
- [Derived] Varsano S, Segev D, Shitrit D. Severe and non-severe asthma in the community: A large electronic database analysis. Respir Med. 2017 Feb;123:131-139. doi: 10.1016/j.rmed.2016.12.017. Epub 2016 Dec 28. PMID 28137489